CLINICAL TRIAL: NCT07184892
Title: Effects of Different Modes of Action Observation Therapy on Swallowing Function After Stroke: a Study Based on fNIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202406-003-1
Record Dates: First submitted 2025-07-20; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; action observation; mirror neurons; Dysphagia; swallowing function
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video swallowing action observation therapy (Active Comparator): On the basis of traditional swallowing training, this group adds video-assisted movement observation therapy, that is, watching swallowing movement videos with sound and then performing simulated swallowing movements.
  Interventions: Behavioral: Video swallowing action observation therapy
- Daily life actual swallowing action observation therapy (Experimental): On the basis of traditional swallowing training, this group adds the practice of observing the real eating and swallowing actions of relatives in actual daily life, and then imitating those swallowing actions.
  Interventions: Behavioral: Daily life actual swallowing movement observation therapy
- Traditional swallowing training (Active Comparator): Routine swallowing function training includes indirect training (basic training) and direct training (feeding training). Indirect training includes but is not limited to training for the muscle strength and range of motion of swallowing muscles, training for inducing swallowing reflexes, breathing training, compensatory swallowing training, and airway protection training. Direct training involves the eating environment, body position, food selection, the amount and speed of each mouthful of food, as well as the compensatory skills commonly used during the eating process.
  Interventions: Behavioral: Traditional swallowing training

INTERVENTIONS:
Behavioral: Daily life actual swallowing movement observation therapy — This group adds the therapy of observing actual swallowing movements in daily life, that is, in real daily life, observing the real eating and swallowing movements of relatives. They select meals that the patient likes or those that are complete in color, aroma and taste and look appetizing. The swallowing movements should be as slow and exaggerated as possible, and a look of savoring and enjoying the food should be shown, so that the patient can better observe the movements of the mouth and larynx during swallowing. Then, the patient imitates the swallowing movements.
  Arms: Daily life actual swallowing action observation therapy
Behavioral: Video swallowing action observation therapy — Video swallowing action observation therapy
  Arms: Video swallowing action observation therapy
Behavioral: Traditional swallowing training — Traditional swallowing training
  Arms: Traditional swallowing training

SUMMARY:
Dysphagia is one of the most common symptoms of stroke patients, which seriously affects the quality of life of patients and delays the progress of rehabilitation. At present, the commonly used clinical swallowing treatment methods can achieve certain therapeutic effects, but the treatment effect of some patients is still not ideal. Therefore, we need to explore more and more effective treatment methods to improve the swallowing function of patients. Action observation therapy, which was developed based on the mirror neuron theory, has been widely used in the rehabilitation of limb motor function, and its therapeutic effect has been verified by a large number of clinical trials. There are few clinical studies on action observation therapy in swallowing function rehabilitation, and most of the current studies use swallowing videos to allow patients to observe actions, and then guide patients to imitate actions. Some studies have found that oral mirror neurons can be formed in the context of familiar environment, people and emotional communication. Therefore, this study proposes a new mode of action observation therapy for dysphagia, that is, to observe the real swallowing movement in actual daily life, in order to better improve the swallowing function of stroke patients with dysphagia.

This study was a single-center, assessor-blinded, randomized controlled study. After enrollment, all patients received swallowing assessment, including scale assessment (WST, FOIS, SSA, BMI, SWAL-QOL, VAS satisfaction survey, KVIQ motor imagery assessment, total oral intake/eating time), neck ultrasound and FNIRS brain function assessment. According to the random number table method, the patients were divided into three groups, A: control group, B: video swallowing movement observation therapy group, C: daily actual swallowing movement observation therapy group. All three groups were given routine swallowing function training. In group B, action observation therapy with video was added, that is, watching a video of swallowing action with sound, and then performing simulated swallowing action. Group C added the actual swallowing movement observation therapy in daily life, that is, in actual daily life, to observe the real eating and swallowing movement of relatives, and then imitate the swallowing movement. The training sessions were 30min each time, once a day, 5 days a week, for a total of 3 weeks. After the treatment, the scale assessment, neck ultrasound and FNIRS brain function assessment were performed again.

ELIGIBILITY:
Inclusion Criteria:

* 1: 1.n accordance with the diagnostic criteria formulated by the Fourth National Academic Conference on Cerebrovascular disease;

  2: 2.Dysphagia was detected by water swallowing test;

  3: 3.First onset, course of disease within 6 months, the condition is stable;

  4: 4.Mini-mental state examination (MMSE) score, literacy >=17 points, primary education >=20 points, secondary education >=24 points, can understand and cooperate with treatment;

  5: 5.Have a certain degree of sitting balance ability, can maintain a sitting position for 30 minutes;

  6: 6.Aged 18-80 years old;

  7: 7.The patient was informed and consented to this study, and the patient's family was informed and trained, and could cooperate with the adjuvant treatment of swallowing movement observation therapy in daily life.

Exclusion Criteria:

* 1: Patients with impaired swallowing function due to other reasons;

  2: Presence of tumors or other lesions in the mouth or throat;

  3: Visual and hearing dysfunction;

  4: The presence of agnosia, apraxia or unilateral neglect;

  5: Severe cognitive impairment and mental and emotional instability can not cooperate with treatment;

  6: Implantation or retention of ferromagnetic metals in the brain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale（FOIS） | Assessment before intervention and 3 weeks after intervention after enrollment.
  This scale is divided into 7 levels in total, which is used to assess the oral feeding ability of the subjects. The higher the level, the better the function.
  Level 1: Unable to take food orally; Level 2: Dependent on tube feeding, able to attempt very small amounts of food or liquids orally; Level 3: Dependent on tube feeding, able to take food or liquids of a single texture orally; Level 4: Completely able to take food of a single texture orally; Level 5: Completely able to take food of multiple textures orally, but requiring special preparation or compensatory measures; Level 6: Completely able to take food orally without special preparation, but with specific food restrictions; Level 7: Completely able to take food orally without any restrictions.

SECONDARY OUTCOMES:
Body Mass Index（BMI） | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  Calculation method for the weight (kg) divided by the square of height (meters).
Through the mouth eating/total time of food intake | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  The time required for patients to eat a given amount of food was recorded.
The neck ultrasound | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  The probe of ultrosound will be placed in the middle of the neck, paralled to the sagittal line. Record the video of participant drinking 1ml water, the distance between hyoid and chin at rest minus distance during hyoid and chin are nerest. Repeated three times, and the mean value is further into analysis.
Score of Water swallow test | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  The patient sat in a upright position and drank 30 ml of warm water. The time required and cough were observed. On a scale of 1-5, the higher the rating, the worse the function.
functional near - infrared spectroscopy（fNIRS） | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  Subjects were calm fNIRS tests 10 ~ 15 minutes rest again, the subjects keep head motionless, resting state, task state data.
Kinesthetic and Visual Imagery Questionnaire（KVIQ) score | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  Subjects were seated and, as requested by the examiner, actually performed motor movements: forward shoulder flexion, finger opposition, forward trunk flexion, hip abduction, and foot tapping. The subject returned to the starting position and imagined the motor action that had actually been performed, but without moving the body. Visual imagery was assessed first, followed by motor imagery. The minimum score of KVIQ-10 is 10 points, and the maximum score is 50 points.
Visual analogue scale（VAS）satisfaction survey score | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  VAS is mainly used to evaluate the degree of pain of patients, and the principle of VAS score can be used for reference when using VAS score for satisfaction investigation. Prepare a 10cm straight line with one end marked "0" to indicate dissatisfaction; The other end is marked with a "10", indicating great satisfaction.
swallowing-quality of life（SWAL-QOL）scale score | Assessments will be conducted after enrollment but before intervention, and three weeks after the intervention.
  A total of 44 questions were classified into 11 dimensions: psychological burden, eating time, appetite, food choice, language communication, fear of eating, mental health, social interaction, fatigue, sleep and swallowing symptoms. Each item is scored by Likert 5-level scoring method (1-5 points correspond to 1-5 points), with a total score of 44 to 220 points. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang C, Li X, Wang H. Application of action observation therapy in stroke rehabilitation: A systematic review. Brain Behav. 2023 Aug;13(8):e3157. doi: 10.1002/brb3.3157. Epub 2023 Jul 21. PMID 37480161
- [Result] Zeng M, Wang Z, Chen X, Shi M, Zhu M, Ma J, Yao Y, Cui Y, Wu H, Shen J, Xie L, Fu J, Gu X. The Effect of Swallowing Action Observation Therapy on Resting fMRI in Stroke Patients with Dysphagia. Neural Plast. 2023 Apr 21;2023:2382980. doi: 10.1155/2023/2382980. eCollection 2023. PMID 37124873
- [Result] Ferrari PF, Gerbella M, Coude G, Rozzi S. Two different mirror neuron networks: The sensorimotor (hand) and limbic (face) pathways. Neuroscience. 2017 Sep 1;358:300-315. doi: 10.1016/j.neuroscience.2017.06.052. Epub 2017 Jul 4. PMID 28687313
- [Result] Jing YH, Lin T, Li WQ, Wu C, Li X, Ding Q, Wu MF, Xu GQ, Lan Y. Comparison of Activation Patterns in Mirror Neurons and the Swallowing Network During Action Observation and Execution: A Task-Based fMRI Study. Front Neurosci. 2020 Aug 21;14:867. doi: 10.3389/fnins.2020.00867. eCollection 2020. PMID 32973431
- See also: Application of action observation therapy in stroke rehabilitation: A systematic review — https://pubmed.ncbi.nlm.nih.gov/37480161/
- See also: The Effect of Swallowing Action Observation Therapy on Resting fMRI in Stroke Patients with Dysphagia — https://pubmed.ncbi.nlm.nih.gov/37124873/
- See also: Two different mirror neuron networks: The sensorimotor (hand) and limbic (face) pathways — https://pubmed.ncbi.nlm.nih.gov/28687313/
- See also: Comparison of Activation Patterns in Mirror Neurons and the Swallowing Network During Action Observation and Execution: A Task-Based fMRI Study — https://pubmed.ncbi.nlm.nih.gov/32973431/